CLINICAL TRIAL: NCT02397668
Title: CorMatrix Cor TRICUSPID ECM Valve Replacement Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corvivo Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-PR-1101 Rev. L
Record Dates: First submitted 2015-03-06; First posted 2015-03-25 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Tricuspid Valve Disease

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, single-arm, Pivotal study of subjects receiving the Cor TRICUSPID ECM Valve or Cor PEDIATRIC Tricuspid ECM Valve
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CorMatrix Cor TRICUSPID ECM Valve (Experimental): Tricuspid valve replacement in patients for the surgical management of tricuspid valve disease, including tricuspid valve disease secondary to congenital heart disease. Enrollment will include up to 60 adults subjects and up to 18 pediatric subjects.
  Interventions: Device: CorMatrix Cor TRICUSPID ECM Valve

INTERVENTIONS:
Device: CorMatrix Cor TRICUSPID ECM Valve — CorMatrix Cor TRICUSPID ECM Valve to replace a diseased tricuspid valve, including tricuspid valve disease secondary to congenital heart disease.
  Other Names: Cor PEDIATRIC Tricuspid ECM Valve

SUMMARY:
The Pivotal Study of the Cor TRICUSPID ECM Valve (or Cor PEDIATRIC Tricuspid ECM Valve). This study follows the EFS and is now to determine the safety and efficacy of the Cormatrix Cor TRICUSPID Valve for any patients requiring surgical replacement of the tricuspid valve.

DETAILED DESCRIPTION:
CorMatrix Cardiovascular, Inc. has developed a device for heart valve replacement, the CorMatrix® Cor ECM® Tricuspid Valve, which can be implanted to replace dysfunctional tricuspid heart valves. This Pivotal Study is being performed to verify the ability to successfully implant the Tricuspid Valve, the clinical safety of the device, and whether the device performs its intended use. The study is a multi-center, prospective, single-arm, Pivotal Study of subjects receiving the Cor TRICUSPID ECM Valve or Cor PEDIATRIC Tricuspid ECM Valve. The study will be conducted at up to 15 sites.

Up to 60 subjects will undergo tricuspid valve replacement (TVR) with the CorMatrix ECM Valve for the surgical management of tricuspid valve disease. The cohort will include up to 60 adult and 18 pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a regurgitant or absent tricuspid valve requiring surgical treatment including those patients having concomitant cardiac procedures
2. Male or female
3. Patient/authorized legal guardian understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provides written informed consent and the pediatric patient (if applicable) provides written assent (if able) prior to procedure
4. Patient/patient's authorized legal guardian is geographically stable (or willing to return for required study follow-up) and understands and is willing to fulfill all of the expected requirements of this clinical protocol
5. Children with congenital disease where the Cor PEDIATRIC Tricuspid ECM Valve would be the physiological right-sided valve

Exclusion Criteria:

1. Tricuspid annulus too small (< 10mm) to accommodate the Cor Tricuspid ECM Valve
2. Left ventricular ejection fraction (LVEF) < 25%
3. Mean pulmonary pressure > 50mm Hg or pulmonary vascular resistance greater than 6 Woods Units
4. Emergency cardiac procedure. An example would be a person requiring resuscitation and in cardiogenic shock. An unscheduled or unplanned emergency surgery
5. Cardiac transplant patient
6. Acute transmural myocardial infarction (MI) within 7 days of enrollment that results in cardiogenic shock
7. Patients with a single ventricle where the Cor Tricuspid ECM Valve would be the systemic AV valve
8. Documented primary coagulopathy or uncorrected platelet disorder, including thrombocytopenia (absolute platelet count <30k). Patient can be enrolled regardless of these parameters if in the opinion of the Investigating Surgeon the coagulopathy can be adequately reversed by transfusions. An example would be the reversal of thrombocytopenia by transfusion of platelets
9. Documented evidence of intrinsic hepatic disease (defined as liver enzyme values (aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin) that are > 5 times the upper limit of reference range within 30 days of enrollment, except in association with acute/reversible decompensation as determined by the Investigator)
10. Documented evidence of significant renal dysfunction (serum creatinine > 4.0mg/dl or GFR< 30 on the modified Schwartz formula)
11. Stroke within 30 days prior to enrollment
12. Major or progressive non-cardiac disease (liver failure, renal failure, cancer (CA)) that has a life expectancy of less than one year
13. Known cancer (cancer-free <1 year; does not include non-metastatic basal cell carcinoma or cervical carcinoma) and/or undergoing treatment including chemotherapy and radiotherapy
14. Hematological disorders (e.g., aplastic anemia) or patients taking bone marrow suppressant drugs
15. Known sensitivity to porcine materials
16. Contraindication to anticoagulation/antiplatelet therapy (aspirin (ASA) and/or Plavix)
17. Patients who are pregnant (method of assessment Investigator's discretion)
18. Patients who are currently enrolled in another investigational study or registry that would directly impact the treatment or outcome of the current study, without CorMatrix written approval

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | 30 days postop
  Device Success and No TV device- or TV procedure-related SAE's

SECONDARY OUTCOMES:
Device Success | 30 day and all follow up time points
  Patient alive with original intended CorMatrix ECM TV in place, No additional surgical or interventional procedures related to the TV, and Intended performance of the TV
Technical Success | within 24 hours
  Exit OR Alive, Successful implant of the single intended CorMatrix ECM TV, No need for additional emergency surgery or re-intervention related to the TV device, Final post-op TTE shows TR < moderate

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Matheny, MD, Study Director — Corvivo Cardiovascular, Inc.
Locations (4):
- United States (4):
  - Springhill Memorial Hospital, Mobile, Alabama
  - St Francis Hospital, Indianapolis, Indiana
  - Medstar, Baltimore, Maryland
  - Cincinnati Children's Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No